CLINICAL TRIAL: NCT01398865
Title: Cerebral Metabolic Correlates of Treatment Response to Escitalopram in Body Dysmorphic Disorder
Brief Title: Escitalopram Neuroimaging Supplement
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sabine Wilhelm, PhD, Massachusetts General Hospital
Other Study IDs: 2008P002032
Record Dates: First submitted 2011-07-15; First posted 2011-07-21 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Body Dysmorphic Disorder
Keywords: BDD
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: PET scan and MRI scan — PET: The PET Scan is manufactured by Siemens and the model is the Exact HR+ .rCMRglu data will be gathered over a 30 minute resting period using a Siemens HR+ PET camera (4.5 mm in-plane and axial resolution). The total time for an individual PET session, will thus be one hour and a half (30 minutes for serum pregnancy test and 30 minute uptake period followed by 30 minutes of scanning).
  MRI: High-resolution scans will be acquired using a Seimens (manufacturer) 1.5T Avonta system at MGH, to be coregistered with subsequently acquired PET images, and used for A) delineation of regions of interest (ROIs), and B) facilitation of optimal transformation to MNI space.

SUMMARY:
The purpose of this study is to find out more about the brain's response to selective serotonin reuptake inhibitor (SSRIs) treatment in people with body dysmorphic disorder (BDD). The investigators will use positron emission tomography (PET) and Magnetic Resonance Imaging (MRI) scans to look at brain activity in people with BDD before and after treatment with an SSRI. The investigators hope that what is learned will allow prediction of whether someone will improve with SSRI treatment.

DETAILED DESCRIPTION:
The investigators have chosen to focus on five regions of interest, namely ACC, OFC, caudate, amygdala and hippocampus. These are brain regions that have been previously associated with obsessive-compulsive, affective, and psychotic phenomena. The investigators will test for correlations between pre-treatment FDG brain images and subsequent SSRI treatment outcome to identify potential predictors of treatment response. Finally, the investigators will compare pre-treatment and post-treatment PET FDG studies as well as MRI studies in BDD subjects to examine changes in these brain regions following treatment. The goals of the proposed research are to use FDG-PET and MRI to identify predictors of treatment response to SSRIs in BDD and to determine changes in rCMRglu in BDD subjects following treatment with SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* male or female.
* from 18-64 years of age.
* right-handed, by virtue of assessment with the Edinburgh Handedness Inventory
* capacity to render informed consent.
* already enrolled in clinical study NCT00149799.
* must be an outpatient with a primary (the condition that is most central to the patient's current distress) psychiatric diagnosis of BDD, as defined by DSM-IV criteria and by a BDD Yale-Brown Obsessive-Compulsive Scale Score greater than or equal to 24.

Exclusion Criteria:

* with serious medical illness or instability for which hospitalization may be likely within four months of entry into the study, or current renal insufficiency or diabetes.
* any pregnant or lactating women or those of childbearing potential not using medically accepted forms of contraception will be excluded. Pregnancy status will be determined by administration of a blood beta-HCG test prior to each PET scan.
* with recent or anticipated radiation exposure, which, combined with the exposure in the present study, will exceed allowable annual limits for the subject
* with a history of hypersensitivity to any component of FDG
* with specific comorbid psychiatric diagnoses (alcohol abuse or dependence within the past 3 months, bipolar disorder, psychosis, organic mental disorder, development disorder, borderline personality disorder, body image concerns accounted for primarily by an eating disorder or weight concerns). If subjects have another comorbid diagnosis, the BDD must be the primary concern.
* MRI- incompatibilities (for example, metal implants, pacemakers)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be 24 subjects with BDD newly enrolled, but not yet treated, in a multi-site (MGH and Rhode Island Hospital) clinical study of escitalopram for BDD (NCT00149799/R01MH072854), Dr. Wilhelm, PI). All BDD subjects will be drawn from this clinical study, in order to best ensure that they have all received a comparable regimen of SSRI treatment. BDD subjects will have been recruited via the BDD Clinic at Massachusetts General Hospital (MGH)/Harvard Medical School and Rhode Island Hospital/Brown Medical School.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
BDD-YBOCS | 9 months
  We will test for correlations between pre-treatment FDG brain images and subsequent SSRI treatment outcome to identify potential predictors of treatment response. Statistical parametric maps will be used to assess the relationship between rCMRglu and subsequent clinical response (expressed as percent change in BDD-YBOCS).

SECONDARY OUTCOMES:
PET FDG and MRI studies | 9 months
  We will compare pre-treatment and post-treatment PET FDG studies as well as MRI studies in BDD subjects to examine changes in these brain regions following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Wilhelm, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- OCD & Related Disorders Clinic, Boston, Massachusetts, United States

REFERENCES:
- See also: Mass General Hospital OCD/BDD clinic website — https://mghocd.org/